CLINICAL TRIAL: NCT00565097
Title: Long-Acting Lanreotide as a Volume Reducing Treatment of Polycystic Livers
Brief Title: Lanreotide as Treatment of Polycystic Livers
Acronym: LOCKCYST
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Ipsen (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMO 2007/010;ABR NL16194.091.0
Record Dates: First submitted 2007-11-28; First posted 2007-11-29 (Estimated); Last update posted 2009-02-17 (Estimated); Status verified 2009-02

CONDITIONS: Polycystic Liver Disease; Hepatomegaly; Liver Diseases; Polycystic Kidney, Autosomal Dominant
Keywords: Polycystic Liver Disease; Autosomal Dominant Polycystic Kidney Disease; Liver cyst; Lanreotide
MeSH Terms: conditions — Polycystic liver disease; Hepatomegaly; Liver Diseases; Polycystic Kidney, Autosomal Dominant | interventions — lanreotide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- 1 (Experimental): Lanreotide
  Interventions: Drug: Lanreotide

INTERVENTIONS:
Drug: Placebo
  Arms: 2
Drug: Lanreotide
  Arms: 1

SUMMARY:
To assess the efficacy of lanreotide in controling total liver volume in patients with polycystic livers this study will be performed. A minimum of 38 patients will be recruited and randomized (1:1) to receive either verum or placebo. Lanreotide is already used in other disease states and found to be safe and non-toxic.

ELIGIBILITY:
Inclusion Criteria:

* 18 yrs-of age
* Multiple cysts > 20
* Cooperating patient
* Is willing and able to comply with the study drug regimen and all other study requirements
* Willingness to give written informed consent

Exclusion Criteria:

* Use of oral anticonceptives or estrogen suppletion
* Females who are pregnant or breast-feeding
* History or other evidence of chronic pulmonary disease associated with functional limitation
* History of severe cardiac disease
* History or other evidence of severe illness or any other conditions which would make the patient, in the opinion of the investigator, unsuitable for the study
* Symptomatic gallstones
* Renal failure requiring hemodialysis

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2007-10

PRIMARY OUTCOMES:
Reduction of total liver volume as determined by CT scan | 6 months

SECONDARY OUTCOMES:
Reduction of liver volume and individual cyst volume on CT scan. | 6 months
Change of kidney volume and individual cyst volume on CT scan | 6 months
Symptom evaluation by (validated) questionnaires | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Joost PH Drenth, MD, PhD, Principal Investigator — Radboud University Medical Center Nijmegen; Loes van Keimpema, MSc, Principal Investigator — Radboud University Medical Center Nijmegen; Frederik Nevens, MD, PhD, Principal Investigator — University Hospital Gasthuisberg, University of Leuven
Locations (2):
- University Hospital Gasthuisberg, Leuven, Belgium
- Radboud University Medical Center, Nijmegen, Netherlands

REFERENCES:
- [Derived] St Pierre K, Cashmore BA, Bolignano D, Zoccali C, Ruospo M, Craig JC, Strippoli GF, Mallett AJ, Green SC, Tunnicliffe DJ. Interventions for preventing the progression of autosomal dominant polycystic kidney disease. Cochrane Database Syst Rev. 2024 Oct 2;10(10):CD010294. doi: 10.1002/14651858.CD010294.pub3. PMID 39356039